CLINICAL TRIAL: NCT02896387
Title: Ex Vivo and in Vitro Assessment of the Pharmacological Properties of Molecule Prima in the Restoration of Physiological Differentiation of Gene p63 Dependant Epithelium
Brief Title: Ability of a Molecule (Prima) to Restore Physiological Differentiation in Epithelium Expressing Gene p63
Acronym: PRIMAculture
Status: Terminated | Type: Observational
Why Stopped: Laboratory change, stem cell circuit stopped
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: EGN_2016_14
Record Dates: First submitted 2016-08-29; First posted 2016-09-12 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Ectodermal Dysplasia
MeSH Terms: conditions — Ectodermal Dysplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ectodermal dysplasia associated with p63 is a rare disease which, in addition to limbic abnormalities, primarily affects the skin and cornea. The most common forms are called Ectrodactyly, Ectodermal dysplasia, palate Key for cleft lip and palate (EEC) and Ankyloblepharon, Ectodermal dysplasia, cleft lip and palate (AEC). Apart from symptomatic treatment, no cure is available. To understand the molecular defects associated with this disease and to identify therapeutic tools, a research team modelized the disease by reprograming EEC and AEC patient fibroblasts in pluripotent stem cells (iPSC), then induced iPSC differentiation in patients and controls epidermal (skin) and limbic (cornea) cells and demonstrated that the mutated cells can reproduce in vitro the abnormalities observed in patients.

P63 gene belongs to the family of p53 gene. The functions of the two proteins are very similar. Data suggest that molecule Prima could reactivate the p63 protein mutated in patients and thus alleviate skin defect healing and limbic regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Patient with genetic pathology of the ocular surface
* Age ≥ 7 years

Exclusion Criteria:

* Agonal glaucoma
* low vision mostly related to retinal pathology
* Pregnant or breast-feeding patient

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with genetic pathology of the ocular surface
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
the differentiation of corneal epithelium by histological observation | baseline
  the differentiation of corneal epithelium by histological observation

CONTACTS AND LOCATIONS:
Overall Officials: Eric GABISON, Principal Investigator — Fondation ophtalmologique de Rothschild
Locations (2):
- France (2):
  - Fondation Opthalmologique A de Rothschild, Paris
  - Hopital Necker, Paris

IPD SHARING:
Plan to Share IPD: Undecided